CLINICAL TRIAL: NCT06931457
Title: Efficacy and Safety of the Application of Pulsed Radiofrequency, Combined With Platelet Rich Plasma, to the Treatment of Idiopathic Glossopharyngeal Neuralgia (GPN): A Study Protocol for a Multi-Center, Prospective, Open-Label, Propensity Score Match Cohort Study
Brief Title: Efficacy and Safety of Pulsed Radiofrequency Combined With Platelet Rich Plasma to Treat Idiopathic Glossopharyngeal Neuralgia (GPN)
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: China-Japan Friendship Hospital (Other); The Second Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Pain Management, Beijing Tiantan Hospital
Other Study IDs: KY 2023-263-03-07
Record Dates: First submitted 2025-04-15; First posted 2025-04-17 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Glossopharyngeal Neuralgia; Pulsed Radiofrequency; Platelet Rich Plasma
MeSH Terms: conditions — Glossopharyngeal Nerve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PRF group: Motor stimulation at 2 Hz, 1.0V will be performed and the negative results indicated that no muscle contraction will be generated. Afterwards, PRF treatment will be performed for 360 seconds. The parameters of PRF application were initiated at the voltage of 45 V, the temperature of 42°C, the pulse rate of 2Hz at the rate of 20 milliseconds.
  The pulse treatment generator will be set to the automatic pulsed radiofrequency mode, with a temperature of 42°C, pulse frequency of 2Hz, pulse width of 20ms and treatment duration of 360s.
- PRF+PRP group: Motor stimulation at 2 Hz, 1.0V will be performed and the negative results indicated that no muscle contraction will be generated. Afterwards, PRF treatment will be performed for 360 seconds. The parameters of PRF application were initiated at the voltage of 45 V, the temperature of 42°C, the pulse rate of 2Hz at the rate of 20 milliseconds.
  The pulse treatment generator will be set to the automatic pulsed radiofrequency mode, with a temperature of 42°C, pulse frequency of 2Hz, pulse width of 20ms and treatment duration of 360s. PRF group will only receive PRF treatment, PRF combined with PRP group, after removing the radiofrequency electrode, 2 ml of LP-PRP mixture will be injected slowly. Additional analgesics will be administered for participants' comfort during and after the procedure. If the patients were not satisfied with the outcome after one month, other treatment options will be available.

SUMMARY:
To investigate the efficacy and safety of the application of PRF combined PRP to the for the treatment of GPN.

ELIGIBILITY:
Inclusion Criteria:

1. age >18 years;
2. diagnosed with idiopathic GPN according to the third International Classification of Headache Disorders (ICHD) classification;
3. patients who failed pharmacotherapy or intolerable side effects of medication;
4. undergoing PRF for GPN;
5. at least 1 month of follow-up recordings.

Exclusion Criteria:

1. Patients with bilateral GPN;
2. Abnormalities in blood measurements, liver and kidney function, blood glucose, coagulation, electrocardiography or chest radiography;
3. Infection at the puncture site;
4. Previous mental illness;
5. Previous history of narcotic drug abuse;
6. Prior anticoagulant or antiplatelet therapy;
7. An implantable pulse generator;
8. Current pregnancy or breast feeding.
9. Patients with incomplete medical records (lack of baseline data or postoperative follow-up data).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suitable participants will be screened at the pain management center of each hospital to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) score | 1day, 3days, 1week, 2weeks, 1month, 3months, 6months, and 1year following the procedure
  Numeric rating scale (NRS) score during resting was used to evaluate pain intensity before and after PRF treatment (0=no pain, 10=intolerable pain)

SECONDARY OUTCOMES:
Barrow Neurological Institute pain scale(BNI score) | 1day, 3days, 1week, 2weeks, 1month, 3months, 6months, and 1year following the procedure
  BNI score during resting was used to evaluate pain relief

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Not yet decided